CLINICAL TRIAL: NCT07071922
Title: User Evaluation of Zelfmoord1813.be and Its Related Websites
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0058
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Suicide Prevention; User Experience
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users of Zelfmoord1813 and related websites: individuals of 16y/o or older who visit(ed) the websites zelfmoord1813.be, werkgroepverder.be, mee-leven.be or komuitjekop.be and understand Dutch
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational one-time questionnaire study without intervention

SUMMARY:
Monitoring the availability and accessibility of suicide prevention information in Flanders remains crucial. In 2022, 1,024 people died by suicide in Flanders, and approximately 10,000 individuals required emergency care following a suicide attempt.

The third Flemish Suicide Prevention Action Plan outlines several strategies aimed at achieving the health objective of reducing the suicide rate by 10% by 2030 compared to 2020.

One of the initiatives under the first Flemish Suicide Prevention action plan was the creation of a central online platform for suicide prevention. This led to the launch of Zelfmoord1813.be at the end of 2013. The platform serves as a central point of access to relevant and scientifically grounded information on suicide prevention in Flanders. It provides immediate crisis support through Zelfmoordlijn 1813, a free and anonymous helpline available via phone, chat, or email. In addition, the site offers resources for professionals, journalists, students, and others seeking information on suicide prevention.

Zelfmoord1813.be targets a broad audience across all age groups . The website is managed by the Flemish Centre of Expertise in Suicide Prevention, the government-appointed partner organization for suicide prevention in Flanders. One of the key responsibilities of the Flemish Centre of Expertise in Suicide Prevention is to regularly assess the use, reach, and relevance of Zelfmoord1813.be, partly through recurring user research.

This user research investigates visitors' reasons for accessing the platform, whether they find what they are looking for, and their satisfaction with the content. The findings help evaluate whether all target groups are being reached effectively and inform future strategies for promotion, content development, and improvements.

A first user study was conducted in 2020. The researchers now aim to repeat this evaluation. In recent years, three affiliated websites have also been launched: WerkgroepVerder.be (for suicide bereavement support), Mee-Leven.be (focused on suicide prevention in the social environment) and KomUitJeKop.be (specifically tailored to men). These websites are also managed by the Flemish Centre of Expertise in Suicide Prevention and will be included in the current study.

The study aims to include 3,000 participants aged 16 and older. Visitors to Zelfmoord1813.be, WerkgroepVerder.be, Mee-Leven.be or KomUitJeKop.be will see a pop-up invitation to participate after 30 seconds, which disappears after 20 seconds. If they click "yes," they are redirected to a Qualtrics page, where they complete a short informed consent and a 5-minute questionnaire before being returned to the original website.

Additionally, a message on each website will read: "We are curious about your opinion of our website. Please take your time to explore the site. When you're ready, you can share your feedback by clicking this link." This allows users to participate after reviewing the content at their own pace.

ELIGIBILITY:
Inclusion Criteria:

* 16 y/o or older
* visit(ed) websites zelfmoord1813.be, mee-leven.be, werkgroepverder.be or komuitjekop.be

Exclusion Criteria:

* /

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Users of Zelfmoord1813.be and its related websites
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the websites | Baseline. Completing the questionnaire will take about 5 minutes
  self-developed questionnaire consisting of 1 multiple-choice question about how they found the website; 1 multiple-choice question on their reason for visiting the website, 1 multiple-choice question on how often they visited the website before; 1 question to rate the website on a scale of 1-10; 2 questions with statements about the website and its content to be rated on 5 point Likert scale; 1 multiple-choice question on the use of AI on websites and 3 open questions for feedback (what was good, what was less good and other suggestions)

OTHER OUTCOMES:
Background characteristics | Baseline. Completing the questionnaire takes up to 5 minutes
  5 questions on background characteristics of participants: age, gender identity, education level, ethnical background, province

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No